CLINICAL TRIAL: NCT03336697
Title: Determining the Microbiota Composition of the Middle Meatus in Parkinson's Disease
Brief Title: Determining the Microbiota Composition of the Middle Meatus in Parkinson's
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Gian Pal, Assistant Professor of Neurological Sciences, Rush University Medical Center
Other Study IDs: 16111609-IRB01
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — we will collect blood samples during the study visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease subjects: Patients with untreated or treated Parkinson's disease ages 45-75.
  Interventions: Diagnostic Test: Nasal swab
- Healthy control subjects: Healthy control subjects ages 45-75.
  Interventions: Diagnostic Test: Nasal swab

INTERVENTIONS:
Diagnostic Test: Nasal swab — a nasal swab will be performed by a trained physician by gently passing of a cotton swab in the nasal passage to get samples from middle meatus. This will be performed under guide of nasal anterior endoscopy to visualize the location of sampling. The cotton swab heads will be placed in sterile tubes and frozen at -80°C until DNA extraction.

SUMMARY:
The exact cause of PD remains unknown, but current theories suggest that it results from a combination of hereditary or genetic factors (i.e. family traits ) and exposure to unknown substances in the environment. The purpose of this study is to investigate whether toxins produced by bacteria that live within the nasal canal (nose) and the intestines of people with PD might have a role in causing the disease. The investigators in this study would like to look at the types of bacteria that live in the nasal canals and intestines of PD subjects and compare them with those of subjects who do not have PD.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with a clinical diagnosis of Parkinson's disease by United Kingdom Parkinson Disease Society Brain Bank criteria will be recruited.

2. Hoehn & Yahr stage 1-3 3. Parkinson's disease symptomatic treatment will be allowed. 4. Subjects with deep brain stimulation are allowed.

Exclusion Criteria:

* 1. Occupation expected to change intestinal flora pattern (e.g. sanitation worker) 2. Treatment with medications that may induce parkinsonism (metoclopramide, typical, or atypical antipsychotic agents) 3. Treatment within 12 weeks with systemic antibiotics 4. Known diagnosis of inflammatory bowel disease 5. Symptomatic organic GI disease other than hemorrhoids and hiatal hernia or abdominal surgeries for symptomatic GI disease such as bowel resection, diverticular surgery, colostomy, etc (subjects with a history of an appendectomy or cholesytectomy for benign disease more than 5 years prior to presentation are allowed).

  6. Symptomatic functional GI disease that significantly impairs intestinal motility such as scleroderma or use of GI motility drugs 7. Acute illness requiring immediate hospitalization 8. Pre-existent organ failure or comorbidities as these may change GI flora:
  1. Liver disease (cirrhosis or persistently abnormal AST or ALT that are 2X> normal);
  2. Kidney disease (creatinine>2.0 mg/dL);
  3. Uncontrolled psychiatric illness;
  4. Clinically important lung disease or heart failure;
  5. HIV disease;
  6. Alcoholism, unreliable drinking history; or consumption of alcohol more than 3 times a week or binge drinking or drinking more than or equal to 3 drinks per occasion;
  7. Transplant recipients;
  8. Diabetes;
  9. Clinically significant dehydration or clinically detectable ascites or peripheral edema or cardiac failure 9. Presence of short bowel syndrome or severe malnutrition with ideal body weight < or = 90% or 10. Estimated survival <1 year and Karnofsky performance status <50%; 11. Use of immunosuppressive medications within 3 months of enrollment 12. Chronic use of diuretics

Ages: 45 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Early to moderate stage Parkinson's disease subjects.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
nasal inflammatory microbiome | 1 year
  For microbiome analysis, in silico community functional predictions will be performed using PICRUSt (Phylogenetic Investigation of Communities by Reconstruction of Unobserved States) and significant differences in Kyoto Encyclopedia of Genes and Genomes (KEGG) ortholog (KO) abundances between groups will be identified. "proinflammatory" and "anti-inflammatory" bacteria taxa will be classified and differences in inflammatory metabolite abundance will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided